CLINICAL TRIAL: NCT00546455
Title: Phase 2 Study of the Assessment of the Insulin Sensitizing Activity of Fenretinide in Subjects With Insulin Resistance With BMI >30Kg/m2, and Liver Inflammation Related to Non-alcoholic Fatty Liver
Brief Title: A Randomized, Double-blind Study of the Effects of Fenretinide Administered in Subjects With Obesity
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was terminated due to expired drug with possibility of re-starting in the future.
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Mario Chojkier, Professor of Medicine, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 061257
Record Dates: First submitted 2007-10-17; First posted 2007-10-19 (Estimated); Results first posted 2021-02-10 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-01

CONDITIONS: Obesity; Insulin Resistance
Keywords: Obesity; insulin resistance
MeSH Terms: conditions — Obesity; Insulin Resistance | interventions — Fenretinide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Subjects in this cohort will be given Fenretinide
  Interventions: Drug: Fenretinide
- B (Placebo Comparator): Subjects in this cohort will be given placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fenretinide — 200 mg/day
  Arms: A
Drug: Placebo — 2 capsules/day
  Arms: B

SUMMARY:
Many metabolic complications of obesity are a consequence of abnormal responses of the liver, muscle, and fat to insulin actions. Fenretinide may improve the effects of insulin, preventing metabolic complications.

ELIGIBILITY:
Inclusion Criteria:

* BMI >30

Exclusion Criteria:

* Diabetes Requiring Medication
* Poorly Controlled Co-Morbidities

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2007-12 (Actual); Primary Completion 2012-01 (Actual); Study Completion 2099-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Mario Chojkier, M.D., Principal Investigator — University of California, San Diego and San Diego VA Healthcare Medical Center
Locations (1):
- University of California at San Diego Hospitals, San Diego, California, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was terminated due to expired drug with possibility of re-starting in the future. For this reason the randomization code has not been broken and the data has not been analyzed and there is no way to report the participant flow.
Groups:
- A- Fenretinide: Subjects in this cohort will be given Fenretinide
  Fenretinide: 200 mg/day
- B-Placebo: Subjects in this cohort will be given placebo.
  Placebo: 2 capsules/day
Period: Overall Study
Arm/Group | A- Fenretinide | B-Placebo
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: This study was terminated due to expired drug with possibility of re-starting in the future. For this reason the randomization code has not been broken and the data has not been analyzed and there is no way to report the baseline population analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | A- Fenretinide | B-Placebo | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Sex: Female, Male
Ethnicity (NIH/OMB)

OUTCOME MEASURES:

1. Primary Outcome: Assessment of the Effect on Insulin Resistance
Description: This study was terminated due to expired drug with possibility of re-starting in the future. For this reason the randomization code has not been broken and the data has not been analyzed and there is no way to report the outcome measures.
Time Frame: 30 days
Population: This study was terminated due to expired drug with possibility of re-starting in the future. For this reason the randomization code has not been broken and the data has not been analyzed and there is no way to report the outcome measures.
Arm/Group | A- Fenretinide | B-Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Assessment of the Biochemical Response in Cholesterol, Glucose and Related Blood Tests.
Description: as for outcome 1
Time Frame: 30 days
Population: as for outcome 1
Arm/Group | A- Fenretinide | B-Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 2 months
Description: This study was terminated due to expired drug with possibility of re-starting in the future. For this reason the randomization code has not been broken and the data has not been analyzed and there is no way to report the adverse events.
Arm/Group | A- Fenretinide | B-Placebo
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
This study was terminated due to expired drug with possibility of re-starting in the future. For this reason the randomization code has not been broken and the data has not been analyzed and there is no way to report the participant flow.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes